CLINICAL TRIAL: NCT05008367
Title: Effect of Dexamethasone as Analgesic Treatment After Total Knee Arthroplasty: Subgroup Analyses of The DEX-2-TKA Randomized Clinical Trial
Brief Title: Effect of Dexamethasone as Analgesic Treatment After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Naestved Hospital (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-KAKG-2021
Record Dates: First submitted 2021-07-13; First posted 2021-08-17 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A (Active Comparator): 24 mg dexamethasone i.v. perioperatively and 24 mg dexamethasone i.v. on the first postoperative day
  Interventions: Drug: Dexamethasone
- Treatment B (Active Comparator): 24 mg dexamethasone i.v. perioperatively and placebo (isotonic saline) i.v. on the first postoperative day
  Interventions: Drug: Dexamethasone; Drug: Isotonic saline
- Placebo (Placebo Comparator): Placebo (isotonic saline) i.v. perioperatively and placebo (isotonic saline) i.v. on the first postoperative day
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Dexamethasone — 24 mg intravenous Dexamethasone (6 ml)
  Arms: Treatment A; Treatment B
Drug: Isotonic saline — 6 ml of isotonic saline
  Arms: Placebo; Treatment B

SUMMARY:
Effect of Dexamethasone as Analgesic Treatment After Total Knee Arthroplasty: Subgroup Analyses of The DEX-2-TKA Randomized Clinical Trial This explorative post-hoc analysis is a substudy of the DEX-2-TKA-trial (NCT03506789) investigating diffefferent subgroups of the patients included in the main trial.

DETAILED DESCRIPTION:
Effect of Dexamethasone as Analgesic Treatment After Total Knee Arthroplasty: Subgroup Analyses of The DEX-2-TKA Randomized Clinical Trial This explorative post-hoc analysis is a substudy of the DEX-2-TKA-trial (NCT03506789) investigating diffefferent subgroups of the patients included in the main trial.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the DEX-2-TKA-trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
Cumulative usage of morphine 0-48 hours postoperatively | Time Frame: 0-48 hours postoperatively
  Morphine administered both as patient-controlled analgesia (PCA) i.v. morphine 0-24 hours and oral morphine on demand 24-48 hours, and any other supplemental morphine administered postoperatively. Consumption in mg

OTHER OUTCOMES:
Subgroup analysis on heterogeneity in intervention effect of age | Time Frame: 0-48 hours postoperatively
  Age (years): > 65 vs. ≤ 65
Subgroup analysis on heterogeneity in intervention effect of sex | Time Frame: 0-48 hours postoperatively
  Sex: male vs. female
Subgroup analysis on heterogeneity in intervention effect of ASA group | Time Frame: 0-48 hours postoperatively
  ASA group classification: I+II vs. III
Subgroup analysis on heterogeneity in intervention effect of preoperative pain at rest | Time Frame: 0-48 hours postoperatively
  VAS (mm): > 30 vs. ≤ 30
Subgroup analysis on heterogeneity in intervention effect of preoperative pain when active | Time Frame: 0-48 hours postoperatively
  VAS (mm): > 30 vs. ≤ 30
Subgroup analysis on heterogeneity in intervention effect of type of anesthesia | Time Frame: 0-48 hours postoperatively
  Type of anesthesia: spinal vs. general Anesthesia+Converted to general anesthesia
Subgroup analysis on heterogeneity in intervention effect of prior daily use (last month) of analgesic medication | Time Frame: 0-48 hours postoperatively
  Prior daily use of paracetamol or NSAID: either parecetamol or NSAID vs. neither parecetamol or NSAID

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Gildhøj Privathospital, Brøndby
  - Bispebjerg Hospital, Copenhagen
  - Sjællands Universitetshospital, Køge, Køge
  - Næstsved Sygehus, Næstved
  - Odense Universitetshospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT05008367/Prot_SAP_000.pdf